CLINICAL TRIAL: NCT06984120
Title: Increased Extravascular Lung Water in Asymptomatic Open-water Swimmers
Status: Recruiting | Type: Observational
Sponsor: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, Maria Hårdstedt, Dr. Maria Hårdstedt, PhD, Specialist Internal Medicine, Dalarna County Council, Sweden
Other Study IDs: SIPE - asymptomatic swimmers
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Edema - Acute; Extravascular Lung Water
Keywords: pulmonary edema; asymptomatic pulmonary edema; swimming induced pulmonary edema; SIPE; pulmonary edema in swimmers; extravascular lung water
MeSH Terms: conditions — Pulmonary Edema | interventions — Oxygen Saturation; Body Temperature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Asymptomatic swimmers: Swimmers (18 years or older) finishing an open-water swimming race during the "Vansbrosimningen" open water swimming event, Sweden, without respiratory symptoms.
  Interventions: Diagnostic Test: Lung ultrasound; Diagnostic Test: Peripheral oxygen saturation; Diagnostic Test: Lung auscultation; Diagnostic Test: Body temperature

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — Four chest regions for both lungs are scanned by lung ultrasound; a positive region defined by the presence of three or more B-line artifacts. Bilateral or unilateral presence of two or more positive regions define positive interstitial syndrome.
Diagnostic Test: Peripheral oxygen saturation — Peripheral oxygen saturation measured by non-invasive pulse oxymetry
Diagnostic Test: Lung auscultation — Clinical auscultation of lungs
Diagnostic Test: Body temperature — Body temperature measured by ear thermometer.

SUMMARY:
Previous studies suggest that increased extravascular lung water might be found in open water swimmers without respiratory symptoms. This study aims to investigate a large number of asymptomatic individuals after an open-water swimming race to assess the prevalence of increased extravascular lung water in asymptomatic open-water swimmers.

DETAILED DESCRIPTION:
Swimming-induced pulmonary edema (SIPE) can occur during open-water swimming. The pathophysiological mechanisms are still partly unknown, but central pooling of blood volume and peripheral vasoconstriction have been suggested as important factors. SIPE is characterized by acute onset of dyspnea and cough, sometimes with excessive sputum and hemoptysis. The condition usually resolves spontaneously, but medical attention can be required in more severe cases.

Previous studies suggest that SIPE is diagnosed by clinical symptoms, decreased peripheral oxygen saturation and signs of pulmonary edema on lung ultrasound. Interestingly, signs of increased extravascular lung water have been found in divers without respiratory symptoms. There are no similar studies regarding open-water swimmers.

This study aims to investigate a large number of swimmers without respiratory symptoms after finishing an open-water swimming race. Prevalence and amount of increased extravascular lung water after swimming will be assessed by lung ultrasound. In addition, individual baseline factors and information about the race associated with increased extravascular lung water will be evaluated. This study will provide better understanding of the pathophysiological mechanism of SIPE.

ELIGIBILITY:
Inclusion Criteria:

* Completion of an open-water swimming race during the "Vansbrosimningen" open-water swimming event
* No respiratory symptoms (dyspnea and/or cough) during or right after the race
* Age ≥ 18 years

Exclusion Criteria:

* Presence of respiratory symptoms (dyspnea and/or cough) during or right after the swimming race
* Declines participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Swimmers of all swimming skills that participate in the open-water swimming event of Vansbrosimningen - a Swedish open-water swimming event that takes place in Vansbro, Sweden
Sampling Method: Non-Probability Sample
Enrollment: 570 (Estimated)
Dates: Start 2025-06-29 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Interstitial syndrome assessed by lung ultrasound (yes/no) | Within 1 hour after termination of swimming
  Four chest regions for both lungs are scanned by lung ultrasound; a positive region defined by the presence of three or more B-line artifacts. Bilateral or unilateral presence of two or more positive regions define positive interstitial syndrome.
Number of regions presenting B-lines on lung ultrasound | Within 1 hour after termination of swimming
  Four chest regions for both lungs are scanned by lung ultrasound; a positive region defined by the presence of three or more B-line artifacts. Assessment of the total number of positive regions.
Absolute number of B-lines on lung ultrasound | Within 1 hour after termination of swimming
  Four chest regions for both lungs are scanned by lung ultrasound; the absolute number of B-lines in each region is counted.

SECONDARY OUTCOMES:
Peripheral oxygen saturation | Within 1 hour after termination of swimming
  Peripheral oxygen saturation measured by non-invasive pulse oxymetry
Presence of crackles on lung auscultation (yes/no) | Within 1 hour after termination of swimming
  Presence of crackles on lung auscultation
Body temperature | Within 1 hour after termination of swimming
  Body temperature measured by ear thermometer
Interstitial syndrome assessed by lung ultrasound (yes/no) | At follow up within 4 hours after termination of swimming
  Four chest regions for both lungs are scanned by lung ultrasound; a positive region defined by the presence of three or more B-line artifacts. Bilateral or unilateral presence of two or more positive regions define positive interstitial syndrome. Performed in individuals with signs of increased extravascular lung water after swimming.
Number of regions presenting B-lines on lung ultrasound | At follow up within 4 hours after termination of swimming
  Four chest regions for both lungs are scanned by lung ultrasound; a positive region defined by the presence of three or more B-line artifacts. Assessment of the total number of positive regions. Performed in individuals with signs of increased extravascular lung water after swimming.
Absolute number of B-lines on lung ultrasound | At follow up within 4 hours after termination of swimming
  Four chest regions for both lungs are scanned by lung ultrasound; the absolute number of B-lines in each region is counted in individuals with sign of increased extravascular lung water after swimming. Performed in individuals with signs of increased extravascular lung water after swimming.
Absolute number of B-lines on lung ultrasound | At baseline 2-4 hours before swimming
  Four chest regions for both lungs are scanned by lung ultrasound; the absolute number of B-lines in each region is counted.
Peripheral oxygen saturation | At baseline 2-4 hours before swimming.
  Peripheral oxygen saturation measured by non-invasive pulse oxymetry
Body temperature | At baseline 2-4 hours before swimming.
  Body temperature measured by ear thermometer
Perceived exertion during swimming | Within 1 hour after termination of swimming
  Perceived exertion during the swimming race measured by "Borg rating of perceived exertion scale". Values on the scale range from a minimum value of 6 (no exertion) to a maximum value of 20 (maximal exertion).

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Center of Clinical Research Dalarna, Falun, Dalarna County
  - Center of Clinical Research Dalarna, Falun

IPD SHARING:
Plan to Share IPD: No